CLINICAL TRIAL: NCT06031558
Title: A Phase III, Open-Label, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of SY-5007, a RET Inhibitor, in Patients With Locally Advanced or Metastatic RET Fusion-positive NSCLC.
Brief Title: Phase III Study of SY-5007, a RET Inhibitor, in Patients With Locally Advanced or Metastatic RET Fusion-positive NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-5007-III-01
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: SY-5007; RET-positive NSCLC; Locally advanced RET-positive NSCLC; Metastatic RET-positive NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SY-5007 (Experimental): SY-5007 will be given orally 160 mg twice daily in 28-day cycle continuously until disease progression, death, unacceptable toxicity, or withdraw consent in this study.
  Interventions: Drug: SY-5007

INTERVENTIONS:
Drug: SY-5007 — a RET selective Inhibitor
  Other Names: SY-5007 tablets

SUMMARY:
This is a phase III, open-label, single-arm, multicenter study designed to evaluate the anti-tumor activity and safety of SY-5007 administered orally to participants with locally advanced or metastatic RET-positive NSCLC.

DETAILED DESCRIPTION:
This study will enroll patients with locally advanced or metastatic RET-positive NSCLC. SY-5007 will be administered orally 160 mg twice daily in 28-day cycle continuously until disease progression, death, unacceptable toxicity, withdrawal of consent, or protocol-specified parameters. This study is designed to evaluate the anti-tumor activity (over response rate [ORR], disease control rate [DCR], duration of response [DOR], progression free survival [PFS] and overall survival [OS]) and safety of SY-5007 in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years old.
2. Histologically or cytologically confirmed diagnosis of locally advanced (with a tumor lesion that cannot be eradicated by surgery or radiotherapy as assessed by the investigators) or metastatic NSCLC.
3. No prior systemic antitumor therapy for locally advanced or metastatic NSCLC (Note: enrollment is permitted in the following 2 situations: 1) received only adjuvant therapy and the end of treatment was ≥ 6 months prior to the first dose; 2) received only radical radiotherapy and the end of treatment was ≥ 6 months prior to the first dose).
4. The patient's tumor tissue or blood sample test result meets 1 of the following two criteria: a. Previous tumor tissue or blood samples are confirmed as RET fusion positive by local laboratory testing. b. If there is no previous RET fusion positive test report, a compliant tumor tissue or blood sample is required to be provided at the central laboratory, using a next-generation sequencing (NGS)-based assay to confirm RET fusion positive.
5. Patients have at least one measurable lesion per RECIST version 1.1. (except for patients with measurable lesions in the brain only) (Note: a lesion that has been treated with radiotherapy or localized therapy is generally not considered a measurable lesion unless there is definitive progression of that lesion).
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
7. Life expectancy of at least 3 months.
8. Patients must have adequate organ function as defined in the below:

   Bone marrow function:

   patients must not have received any blood products, hematopoietic cell growth factors or other blood medications for at least 7 days prior to the first dose, and have a blood count: absolute neutrophil count (ANC) ≥ 1.5 x 10^9 /L, platelet (PLT) count ≥ 75 x 10^9 /L, and hemoglobin (Hb) ≥ 90 g/L;

   Liver function:

   total bilirubin (TBIL) ≤ 1.5 times upper limit of normal (ULN) and both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN in the absence of liver metastases; in the presence of liver metastases, both AST and ALT ≤ 5.0 times ULN and TBIL ≤ 3 times ULN;

   Renal function:

   creatinine clearance (Ccr) ≥ 50 mL/min.

   Coagulation function:

   prothrombin time (PT) or International Normalized Ratio (INR) ≤ 1.5 times ULN.
9. Patients can swallow the drug orally and are able to comply with follow-up visit requirements.
10. Male and female patients of childbearing potential must be willing to abstain completely or agree to use an appropriate method of contraception for the duration of the study and for at least 3 months after the last dose of study medication.

Exclusion Criteria:

1. Patients carried known major driver genetic alterations other than RET. e.g. EGFR, MET, ALK, ROS1, NTRK, BRAF V600, KRAS G12C, etc. (If a patient has a co-mutation, discuss with the investigators whether enrollment is possible).
2. History of allergy to any components or excipients of SY-5007 tablets.
3. Patients with malignancies other than NSCLC treated in this study (except: malignancies that are cured and have not recurred within 2 years prior to study entry; completely resected basal cell and squamous cell skin cancer; completely resected carcinoma in situ of the cervix or breast).
4. Patient has clinically symptomatic primary central nervous system (CNS) tumor, symptomatic CNS metastases, molluscum contagiosum, or untreated spinal cord compression; exclusion: patient has stable CNS disease (no evidence of progression as determined by imaging for at least 4 weeks prior to the first dose and all neurological symptoms have returned to baseline levels), no evidence of new or enlarging brain metastases, and has not had CNS surgery or radiotherapy within 4 weeks prior to the first dose, has not undergone stereotactic radiosurgery within 2 weeks, and has discontinued or stabilized steroid dosing within 2 weeks.
5. Comorbidities of the following symptoms or conditions prior to the first dose that remain poorly controlled with optimal therapy:

   active uncontrolled systemic bacterial, viral, or fungal infections; pleural, abdominal, or pericardial effusions that are poorly controlled with interventions (e.g., drainage) (poorly controlled is defined as growth that is significant and symptomatic within 2 weeks of fluid collection and requires re-puncturing or other interventions); poorly controlled diabetes mellitus [fasting blood glucose ≥ 10 mmol/L and/or glycated hemoglobin (HbA1c) ≥ 8%]; uncontrolled symptomatic hyperthyroidism or hypothyroidism as assessed by the investigators; uncontrolled electrolyte disorders (e.g., hyper/hypocalcemia, hyper/hypomagnesemia, hyper/hypokalemia) as assessed by the investigators; clinically significant severe gastrointestinal disorders as assessed by the investigators, including active ulcerative colitis Crohn's disease, peptic ulcers, or previous surgical procedures that may have significantly interfered with the absorption of the drug.
6. Presence of serious cardiovascular disease/abnormalities as indicated by any of the following:

   a QTcF > 470 msec (females) or > 450 msec (males) using the Fridericia formula for heart rate correction at screening, (If drug-induced prolongation of the QTcF is suspected, it is assessed by the investigators to be safe and manageable and may be corrected with medication and then enrolled.); left ventricular ejection fraction (LVEF) < 45%; myocardial infarction or unstable angina pectoris or clinically significant uncontrolled arrhythmia within 6 months prior to the first dose of the drug, including bradyarrhythmias (e.g., type II second or third-degree heart block) that may result in prolongation of the QTcF; classified as class III or IV according to New York Heart Association (NYHA) criteria Congestive heart failure; poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg), history of unstable hypertension, or history of poor compliance with antihypertensive therapy.
7. Presence of active viral infection or history of:

   Hepatitis B (Hepatitis B surface antigen [HBsAg] positive with HBV DNA test > 2 x 10^3 IU/mL, eligible for enrollment if re-tested to less than 2 x 10^3 IU/mL with regular antiviral therapy); positive test for Human Immunodeficiency Virus (HIV) at screening or a known history of other immune deficient disorders; a history of prior organ transplantation, hematopoietic stem cell or bone marrow transplantation therapy.
8. Presence of other lung diseases that require systemic treatment or are serious, such as active tuberculosis, interstitial lung disease, etc., which in the opinion of the investigators may influence the interpretation of the study results or put the patient at high risk.
9. Patients who had used or were unable to discontinue the following potent inhibitors or inducers of CYP3A4 during the study period within 2 weeks prior to the first dose. CYP3A4 potent inhibitors: atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, vinpocetine, voriconazole; and CYP3A4 potent inducers: carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin.
10. Palliative radiotherapy within 1 week prior to the first dose, or any lung radiotherapy with more than 30 Gy of radiation within 6 months prior to the first dose.
11. Major surgical procedure (except central venous catheterization, tumor puncture biopsy, and gastric tube placement) or significant trauma within 4 weeks prior to the first dose.
12. Participation in another clinical trial within 4 weeks prior to the first dose (note: except for those who are not using the investigational drug or investigational medical device; or those who have discontinued treatment from another clinical trial and are only being followed for subsequent survival) or are planning to participate in another clinical trial during the study period.
13. Serious arterial/venous thrombotic event within 1 year prior to the first dose, such as cerebrovascular accident, deep vein thrombosis, pulmonary embolism, or bleeding tendency within 30 days prior to the first dose, or risk of gastrointestinal bleeding as judged by the investigators.
14. Female patients who are pregnant or breastfeeding.
15. Any other conditions that, in the opinion of the investigators, makes participation in this clinical trial inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of ORR by independent review committee (IRC). | Tumor scans performed at baseline then every 8 weeks up to 1 year, then every 12 weeks thereafter; up to 3 years.
  Defined as the number (%) of patients with measurable disease with response of complete response (CR) or partial response (PR) assessed by IRC according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
ORR as assessed by investigators. | Up to 3 years.
  Defined as the number (%) of patients with measurable disease with response of CR or PR assessed by investigators according to RECIST version 1.1.
DCR as assessed by investigators and IRC. | Up to 3 years.
  Defined as the number (%) of patients who have a best overall response of CR or PR or stable disease (SD) according to RECIST 1.1.
PFS as assessed by investigators and IRC. | Up to 3 years.
  PFS is defined as the time from the date of randomization to progression of tumor as assessed by investigators or death from any cause on study.
Time to response (TTR) as assessed by investigators and IRC. | Up to 3 years.
  TTR is defined as the time from the date of randomization to the first response of CR or PR.
DoR as assessed by investigators and IRC. | Up to 3 years.
  DoR is defined as the time from first response until disease progression or death, whichever occurs first.
Overall survival (OS). | Up to 3 years.
  OS is defined as the time from the date of randomization until death due to any cause.
Incidence of adverse events (AEs) and serious adverse events (SAEs). | From the screening period to 28 days after treatment completion, up to a maximum of approximately 3 years.
  AEs are graded according to CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China